CLINICAL TRIAL: NCT04393519
Title: Non-invasive Evaluation of Prognostic Parameters for Patients With Transjugular Intrahepatic Portosystemic Shunt (TIPS) Using a Structured Follow up Protocol 2
Brief Title: Non-invasive Evaluation Program for TIPS and Follow Up Network 2 (NEPTUN2)
Acronym: NEPTUN2
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Michael Praktiknjo, Principal Investigator, University Hospital, Bonn
Other Study IDs: NEPTUN2
Record Dates: First submitted 2020-05-12; First posted 2020-05-19 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Portal Hypertension
Keywords: transjugular intrahepatic portosystemic shunt (TIPS); non-invasive assessments; Transthoracic echocardiography (TTE) with Speckle-tracking; Computer tomography scan (CT-scan); Magnetic resonance imaging (MRI); Circulating biomarkers; Electroencephalography (EEG); Elastography
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, stool, ascites, DNA, PBMC, Buffi coat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective: Prospective cohort that received TIPS from 05/12/2020 onwards
  Interventions: Device: TIPS procedure

INTERVENTIONS:
Device: TIPS procedure — Implantation of TIPS for portal hypertension

SUMMARY:
Evaluation of non-invasive prognostic parameters in patients receiving transjugular intrahepatic portosystemic shunt (TIPS) for complications of portal hypertension. Patients are cared according to the local standardized follow up program. Clinical and laboratory data from standard patient care are evaluated for potential prognostic value.

DETAILED DESCRIPTION:
NEPTUN consists of liver cirrhosis receiving transjugular intrahepatic portosystemic shunt (TIPS) at the Department of Internal Medicine I, University of Bonn, Germany and receiving a structured routine evaluation and follow up program. The diagnosis of cirrhosis was based on clinical, hemodynamic and biochemical parameters, and ultrasound and/or biopsy criteria.

ELIGIBILITY:
Inclusion Criteria:

* Insertion of TIPS according to guidelines

Exclusion Criteria:

* Contraindication for TIPS

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients receiving TIPS according to guidelines
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-05-12 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | up to 10 years
  death, liver transplantation

SECONDARY OUTCOMES:
Ascites | up to 10 years
  Evaluation of amount of ascites according to the Child-Score (0=none;1=moderate/treatable; 2=severe/refractory)
Hepatic Encephalopathy (HE) | up to 10 years
  Evaluation of the grade according to the West Haven Criteria (Grade 0 (no HE) - Grade 4 (hepatic coma))
Variceal Bleeding | up to 10 years
  Assessment of presence of variceal bleeding
Liver Failure | up to 10 years
  defined as Bilirubin level ≥ 12mg/dl
Acute-on-Chronic Liver Failure (ACLF) | up to 10 years
  Presence of ACLF according to the EASL-Chronic liver Failure Consortium (CLIF)-criteria
Organ Failures | up to 10 years
  Assessment of Organ failures according to CLIF-Sequential Organ Failure Assessment (SOFA) Score (Score 6 (best) to 18 (worst))
Kidney Failure | up to 10 years
  Assessment of AKI according to KDIGO definition
Sarcopenia | up to 10 years
  Assessment of sarcopenia according to EASL-guideline definition
post-surgical survival | up to 10 years
  Assessment of post-surgical survival

CONTACTS AND LOCATIONS:
Overall Officials: Michael Praktiknjo, MD, Principal Investigator — University of Bonn
Locations (1):
- University Hospital Bonn, Bonn, Germany

REFERENCES:
- [Derived] Heger LA, Chang J, Rohrer C, Reincke M, Eyth A, Sturm L, Schultheiss M, Maier A, Meyer C, Jansen C, Graf K, Ozturk C, Schneider F, Trebicka J, Westermann D, Thimme R, Grundmann S, Praktiknjo M, Bettinger D. Right Ventricular Contractility Predicts Clearance of Ascites After Transjugular Intrahepatic Portosystemic Shunt. Liver Int. 2025 Dec;45(12):e70422. doi: 10.1111/liv.70422. PMID 41204773